CLINICAL TRIAL: NCT03073915
Title: The Risk for VTE Among Patients in the Medical Wards - Prospective Observational Study.
Brief Title: Evaluation of the Risk of VTE Among Patients Hospitalized in Non-surgical Departments
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0090-08-HMO
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients hospitalized in internal wards are at risk for VTE. The current guidelines recommend the use of thromboprophylaxis for 7-10 days among patients who are at increased risk for VTE. Yet several retrospective studies have shown that the compliance with this guideline is low. Physicians are often reluctant to administer LMWH to their fragile patients mainly because they are not convince that the risk associated with such therapy is greater than the risk for VTE.

In the current study, data concerning the use of thromboprophylaxis among patients admitted to the medical wards will be collected. The occurrence of bleeding or thrombotic event will be evaluated prospectively.

DETAILED DESCRIPTION:
Data concerning the use of LMWH among patients admitted to the medical wards at the Hadassah University Hospital will be collected prospectively from the electronic medical records. The occurrence of bleeding episodes or thrombotic events will be followed for the next 90 days following discharge from the hospital.

The percent of patients actually treated by LMWH among patients entitled for such therapy according to the most updated international guidelines will be evaluated. The risk of minor and major bleeding will be compared among those given thromboprophylaxis and those who were not treated. Similar comparison will be made for thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical wards at the Hadassah University Hospital

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the medical wards at the Hadassah University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Thrombosis | 90 days
  Rate of thrombotic events within 90 days following discharge
Bleeding | 90 days
  Rate of minor and major bleeding episodes within 90 days following discharge
Compliance | 90 days
  Rate of compliance with ACCP guidelines concerning thromboprophylaxis of non-surgical patients.

IPD SHARING:
Plan to Share IPD: Undecided